CLINICAL TRIAL: NCT04471194
Title: Multilevel Intervention Based on CRC and Cervical Cancer Self-screening in Rural, Segregated Areas
Brief Title: Multilevel Intervention Based on Colorectal Cancer (CRC) and Cervical Cancer Self-screening in Rural, Segregated Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer L. Moss, PhD, Assistant Professor, Department of Family and Community Medicine / Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STUDY00015480; K22CA225705-01A1 (NIH)
Record Dates: First submitted 2020-07-04; First posted 2020-07-15 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer Screening; Cervical Cancer Screening
Keywords: Environmental barriers to cancer screening; Person-level barriers to cancer screening
MeSH Terms: interventions — Occult Blood

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Self-Sampling Intervention (Experimental): Participants in this group will receive cervical and colorectal cancer self-sampling kits, instructions for completing the self-sampling kits, and educational materials about cervical and colorectal cancer.
  Interventions: Diagnostic Test: Self-sampling HPV test; Diagnostic Test: Fecal occult blood test
- Control (No Intervention): Participants in this group will receive a standardized letter informing them that they are out-of-date for both cervical and colorectal cancer screenings and should schedule an appointment with their provider to receive these screenings.

INTERVENTIONS:
Diagnostic Test: Self-sampling HPV test — Tests for human papillomavirus from cervical cell sample
  Other Names: Evalyn® Brush
  Arms: Self-Sampling Intervention
Diagnostic Test: Fecal occult blood test — Tests for human hemoglobin from blood in fecal samples
  Other Names: InSure® test
  Arms: Self-Sampling Intervention

SUMMARY:
In this study, the investigators will deliver self-sampling human papillomavirus (HPV) tests and fecal immunochemical test (FIT) kits, as well as adapted cancer screening educational materials, by mail to 110 women who are out-of-date for both cervical and colorectal cancer screenings, recruited through federally qualified health centers (FQHCs) in rural, segregated counties of Pennsylvania.

The hypothesis is that delivering self-sampling HPV tests and FIT, as well as adapted educational materials, to women in rural, segregated areas could help increase cancer screening, reduce geographic cancer disparities, and improve public health.

DETAILED DESCRIPTION:
In this study, the investigators will deliver self-sampling human papillomavirus (HPV) tests and fecal immunochemical test (FIT) kits, as well as adapted cancer screening educational materials, by mail to 110 women who are out-of-date for both cervical and colorectal cancer screenings, recruited through federally qualified health centers (FQHCs) in rural, segregated counties of Pennsylvania. A control group of 110 women, also recruited through FQHCs in rural, segregated counties of Pennsylvania, will be used for comparison; these women will receive standard-of-care reminders for cancer screening and complete the baseline and follow-up surveys.

The hypothesis is that delivering self-sampling HPV tests and FIT, as well as adapted educational materials, to women in rural, segregated areas could help increase cancer screening, reduce geographic cancer disparities, and improve public health.

ELIGIBILITY:
Inclusion Criteria:

* lives in rural, segregated county of Pennsylvania
* able to speak, read, and communicate well in English
* out of date for both cervical and colorectal cancer screening

Exclusion Criteria:

* has had a partial or complete hysterectomy
* has a family history of colorectal cancer
* has a personal history of cervical or colorectal cancer
* persons who are cognitively impaired
* persons who are incarcerated

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Moss, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The research team sent 3436 patients invitations to participate in the study. 200 patients responded. Of the 200 respondents that were contacted for follow-up: 62 were unreachable, 90 were ineligible to participate due to having a hysterectomy, and 48 were enrolled.
Period: Overall Study
Arm/Group | Self-Sampling Intervention | Control
Started | 24 | 24
Completed | 21 | 21
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Sampling Intervention | Control | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 47
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (4.4) | 56 (4.3) | 56 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 20 | 40
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
household income [Count of Participants; unit: Participants]
  < $50,000 | 17 | 15 | 32
  $50,000+ | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentage of Participants Who Completed Any Cervical PLUS Colorectal Cancer Screening Tests
Description: Difference in percentage of participants who self-report having had cervical cancer screening PLUS having had colorectal cancer screening (all modalities) by the end of the study period between the two arms.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Sampling Intervention | Control
Number analyzed (Participants) | 24 | 24
Participants | 18 | 1

2. Secondary Outcome: Difference in Percentage of Participants Who Completed At-home Cervical PLUS Colorectal Cancer Screening Tests
Description: Difference in percentage of participants who completed at-home cervical cancer screening test PLUS completed at-home colorectal cancer screening test by the end of the study period between the two arms.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Sampling Intervention | Control
Number analyzed (Participants) | 24 | 24
Participants | 17 | 0

ADVERSE EVENTS:
Time Frame: 10 weeks (from the time of consent until the completion of the follow-up survey)
Arm/Group | Self-Sampling Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
Low recruitment of minorities; Lack of sufficient power in statistical analyses; Use of cervical cancer screening methods unapproved by the FDA, Use of self-report for primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT04471194/Prot_SAP_002.pdf
  • Informed Consent Form (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04471194/ICF_001.pdf